CLINICAL TRIAL: NCT06892743
Title: Analgesic Efficacy of Ultrasound-guided External Oblique Intercostal Plane Block Versus Posterior Transversus Abdominis Plane Block in Patients Undergoing Open Nephrectomy: A Randomized Double-blinded Comparative Study
Brief Title: Analgesic Efficacy of Ultrasound-guided External Oblique Intercostal Plane Block Versus Posterior Transversus Abdominis Plane Block in Patients Undergoing Open Nephrectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Abeer Ahmed, MD, Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MS-389-2024
Record Dates: First submitted 2025-03-09; First posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EOIPB-Group (Active Comparator)
  Interventions: Procedure: US-guided external oblique intercostal plane block (EOIPB)
- Posterior TAP - Group (Active Comparator)
  Interventions: Procedure: US-guided external oblique intercostal plane block (EOIPB)

INTERVENTIONS:
Procedure: US-guided external oblique intercostal plane block (EOIPB) — US Guided external oblique intercostal plane block (EOIPB) or Posterior TAP Block:
  Other Names: US Guided Posterior TAP Block:

SUMMARY:
Renal cell carcinoma (RCC) accounts for 2-3% of all cancers and is a common malignancy of the genitourinary tract. Open nephrectomy, performed through midline, subcostal, or flank incisions, remains a standard treatment but often results in significant postoperative pain, leading to respiratory muscle dysfunction, increased pulmonary complications, and prolonged hospital stays.

Acute surgical pain arises from inflammatory responses, activation of spinal pain pathways, and muscle spasms. While postoperative pain typically improves during recovery, some patients develop chronic postsurgical pain (CPSP), lasting at least two months postoperatively.

Opioids and epidural analgesia are commonly used for pain control, but their side effects and invasiveness necessitate safer, effective alternatives. Ultrasound (US)-guided peripheral nerve and field blocks have become integral to multimodal analgesia. One such technique, the **external oblique intercostal plane block (EOIPB)**, was introduced as a modification of fascial plane blocks, targeting anterior and lateral cutaneous nerves (T6-T10). EOIPB offers advantages over quadratus lumborum block (QLB) and erector spinae plane block (ESPB) by being performed in the supine position and providing superior midline analgesia compared to serratus intercostal plane block (SIPB).

Similarly, the transversus abdominis plane (TAP) block, particularly the posterior approach, delivers analgesia from T7 to T12 by anesthetizing anterior and lateral cutaneous nerve branches. While case series suggest EOIPB may be effective for post-nephrectomy pain, comparative studies between EOIPB and posterior TAP block in open nephrectomy:

Aim of the Study:

To evaluate the postoperative analgesic effects of posterior transversus abdominis plane (TAP) block and external oblique intercostal plane block (EOIPB) in patients undergoing open nephrectomy under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients whom diagnosed as having renal carcinoma and scheduled for open nephrectomy under general anesthesia.
* ASA class II- III.
* Age ≥ 18 and ≤ 65 years.
* Body mass index (BMI) less than 40kg/m2.

Exclusion Criteria:

* 1. Patient refusal. 2. Hepatic and renal insufficiency. 3. Unstable cardiovascular or pulmonary disease. 4. History of psychiatric and cognitive disorders. 5. Patients with known sensitivity or contraindications to the drug used. 6. Patients on regular opioid consumption.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Postoperative morphine consumption (mg) in the first 24 hrs . | Time elapsed from the end of the block procedure till the end of the 24 hours postoperatively

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Abeer Ahmed Mohamed, Maadi, Cairo Governorate
  - Kasr Alainy Faculty of Medicine - Cairo university, Cairo